CLINICAL TRIAL: NCT04287179
Title: Effect and Safety of Two Different Dose-escalation Regimens for Once-weekly Semaglutide s.c. in Subjects With Type 2 Diabetes Mellitus Previously Treated With GLP-1 RAs
Brief Title: SUSTAIN SWITCH: A Research Study to Compare Two Dose Schedules of Semaglutide Taken Once Weekly in People With Type 2 Diabetes
Acronym: SUSTAIN SWITCH
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: COVID19 impact on this trial was evaluated and a delay of at least 6-9 months was expected. In parallel, the development of a new type of pen injector, which was an important part of the trial, was ceased and thus this trial was cancelled.
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-4650; U1111-1242-5426 (Other: World Health Organization (WHO)); 2019-004234-42 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide 0.50 mg (Experimental): Once-weekly semaglutide administered subcutaneously (s.c., under the skin) with or without oral antidiabetics (OADs). Start dose 0.50 mg.
  Interventions: Drug: Semaglutide
- Semaglutide 0.25 mg (Active Comparator): Once-weekly semaglutide administered subcutaneously (s.c., under the skin) with or without oral antidiabetics (OADs). Start dose 0.25 mg.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Dose gradually increased over 12 weeks to 2.0 mg, followed by a 5 week maintenance period.

SUMMARY:
This study compares the effect and safety of 2 dose schedules for semaglutide (study medicine) in people with type 2 diabetes previously treated with a diabetes medicine similar to semaglutide. The study will also evaluate the use of a new pen-injector for semaglutide used to inject medicine under the skin, at a new dose of 2 mg. People taking part in the study will take this medicine together with their current diabetes tablets other than semaglutide. Participants will either get a start dose of 0.25 mg semaglutide or 0.50 mg semaglutide, and the dose will be gradually increased to 2.0 mg semaglutide - which treatment is decided by chance. Participants will inject semaglutide under the skin once a week, any time of the day. When the dose reaches 2.0 mg semaglutide, participants will inject the medicine with a new type of pen-injector. The study will last for about 24 weeks. Participants will have 9 visits and 1 phone call with the study doctor. At 9 visits participants will have blood taken and at 2 visits they will have eye examination done. Women cannot take part if pregnant, breast-feeding or planning to become pregnant during the study period. Women who are able to get pregnant will be checked 10 times for pregnancy via urine tests.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older at the time of signing informed consent.
* Diagnosed with type 2 diabetes mellitus at least 180 days prior to the day of screening.
* The need and willingness to change prior GLP-1 RA treatment to once-weekly semaglutide s.c., as assessed by the investigator.
* HbA1c of 6.5-10% (48-86 mmol/mol) (both inclusive).
* Treatment with any therapeutic dose of GLP-1 RA other than once-weekly semaglutide s.c., as defined in the local label, with or without OADs (metformin, DPP-4 inhibitor, SU, glinide, thiazolidinedione, SGLT-2 inhibitor or alpha-glucosidase inhibitor). All doses of antidiabetic treatments should have been stable for at least 90 days prior to the day of the screening, at investigator's discretion.

Exclusion Criteria:

* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within the past 90 days prior to the day of screening. However, short term insulin treatment for a maximum of 14 days prior to the day of screening is allowed, as is prior insulin treatment for gestational diabetes.
* Renal impairment measured as estimated glomerular filtration rate (eGFR) value of less than 30 mL/min/1.73 m2 according to Chronic Kidney Disease Epidemiology Collaboration (CKDEPI) creatinine equation as defined by KDIGO 2012 classification.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-11-16 (Estimated); Study Completion 2021-01-25 (Estimated)

PRIMARY OUTCOMES:
Change in glycosylated haemoglobin (HbA1c) | From baseline (week 0) to week 12
  Percent-point

SECONDARY OUTCOMES:
Change in fasting plasma glucose | From baseline (week 0) to week 12
  mmol/L
Change in body weight | From baseline (week 0) to week 12
  Kg
Number of treatment emergent adverse events (TEAEs) | From baseline (week 0) to week 12
  Count
Number of treatment emergent gastrointestinal adverse events | From baseline (week 0) to week 12
  Count
Number of treatment emergent severe or blood glucose confirmed symptomatic hypoglycaemic episodes | From baseline (week 0) to week 12
  Count
Change in pulse rate | From baseline (week 0) to week 12
  Beats per minute (bpm)
Number of treatment emergent adverse events (TEAEs) | From week 12 to week 17
  Count

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor & Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (24):
- United States (14):
  - Novo Nordisk Investigational Site, Buena Park, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, San Jose, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
- Austria (3):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Stockerau
  - Novo Nordisk Investigational Site, Vienna
- Finland (5):
  - Novo Nordisk Investigational Site, Jyväskylä
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Lahti
  - Novo Nordisk Investigational Site, Raisio
  - Novo Nordisk Investigational Site, Seinäjoki
- Sweden (2):
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Malmo

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials. com
URL: http://novonordisk-trials.com